CLINICAL TRIAL: NCT03361631
Title: Intracavernous Injection of Autologous Mesenchymal Stem Cells in the Curative Treatment of Erectile Dysfunction Resistant to Oral Treatment in Patients With Type I Diabetes: Dose Escalation Trial
Brief Title: Intracavernous Injection of Autologous Mesenchymal Stem Cells in the Treatment of Erectile Dysfunction Resistant to Oral Treatment in Patients With Type I Diabetes
Acronym: MESERIC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHRCI2016/MESERIC-EL OSTA/NK
Record Dates: First submitted 2017-11-22; First posted 2017-12-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-11

CONDITIONS: Erectile Dysfunction; Stem Cells; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Erectile Dysfunction; Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- arm treated with MSC (Experimental): * Type 1 diabetic man
  * Aged from 18 to 50 years
  * Having a diabetes evolving for at least 10 years
  * Presenting at least one severe manifestation of microangiopathy, with or without dysautonomia: diabetic retinopathy, diabetic or vascular nephropathy, diabetic neuropathy, diabetic foot
  * Presenting an erectile dysfunction refractory to oral treatment (sildenafil, tadalafil ...)
  * IIEF-5 score less than or equal to 10
  Interventions: Drug: Autologous Bone Marrow derived Mesenchymal Stem Cells

INTERVENTIONS:
Drug: Autologous Bone Marrow derived Mesenchymal Stem Cells — Information visit (time 1) Inclusion visit (time 2) Bone marrow extraction (time 3) Treatment and culture of MSC (time 4) Intra-cavernosal injection of autologous MSC (time 5) Follow-up 1 (time 6): control / tolerance visit (andrological clinical examination, EHS and and IIEF-5), 2 weeks after injection; Follow-up 2 (time 7): 12-week evaluation of treatment response: andrological clinical examination, IIEF-5 and EHS score determination & Pharmaco-Doppler; Follow-up 3 (time 8): 24-week evaluation of the response to treatment: andrological clinical examination, determination of IIEF-5 and EHS scores & Pharmaco-Doppler

SUMMARY:
Diabetes is a major concern in public health because of its high frequency and its negative consequences. Erectile dysfunction (ED) is present, regardless of age, in 50 to 75% of men with diabetes. It is related to endothelial dysfunction and a decrease in smooth muscle and nerve cells. In type 1 diabetic patients, ED is part of the chronic complications of microangiopathy. Current therapies are exclusively symptomatic with moderate efficacy, estimated between 44 and 56%. The administration of culture-grown medullary mesenchymal stem cells (MSCs) would be a curative treatment and have the advantage of being single injection.

However, the data in the literature do not allow to define the optimal dose of MSC in this indication. In addition, the feasibility of this procedure is not known at present.

The aim of this study is to evaluate the tolerance and the efficacy of intracavernous injection of autologous MSC (bone marrow-derived MSCs) administered in a 4-dose-escalating design in patients from 18 to 50 years old with complicated type 1 diabetes mellitus and erectile dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetic man
* Aged from 18 to 50 years
* Having a diabetes evolving for at least 10 years
* Presenting at least one severe manifestation of microangiopathy, with or without dysautonomia: diabetic retinopathy, diabetic or vascular nephropathy, diabetic neuropathy, diabetic foot
* Presenting an erectile dysfunction refractory to oral treatment (sildenafil, tadalafil ...)
* IIEF-5 score less than or equal to 10

Exclusion Criteria:

* Any intercurrent event that does not allow the injection of aMSC
* Violation of the protocol by self erectile dysfunction medication
* Withdrawal of the protocol

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Estimated)
Dates: Start 2018-06-30 (Estimated); Primary Completion 2018-07-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the occurrence of clinical adverse event (tolerance) to intracavernous injection of autologous MSC in patients 18 to 50 years of age with complicated type 1 diabetes mellitus with erectile dysfunction refractory to oral treatment. | within 2 weeks after the injection of CSMa
  Occurrence within 2 weeks after the injection of CSMa at the expected dose (10.106, 20.106, 30.106 and 40.106) of a clinical adverse event: thrombosis (s) of the cavernous body, subcutaneous hematoma, induration of the cavernous body , local inflammatory reaction (redness, pain), general effects: fever, chills

SECONDARY OUTCOMES:
Evaluation of the efficacy of autologous MSC intracavernous injections at different doses with evaluation of the clinical score IIEF-5 (International Index of Erectile Function-5) | 12 and 24 weeks after injection
  Simplified Scale IIEF-5 with 5 questions (total score between 1 to 25)
Evaluation of the efficacy of autologous MSC intracavernous injections at different doses with evaluation of the EHS score | 12 and 24 weeks after injection
Evaluation of the efficacy of autologous MSC intracavernous injections at different doses with evaluation of arterial insufficiency | 12 and 24 weeks after injection
Evaluation of the efficacy of autologous MSC intracavernous injections at different doses with evaluation of venous insufficiency (venous leakage) | 12 and 24 weeks after injection
Evaluation of the feasibility of the autologous MSC intracavernous injection protocol by the number of bone marrow extraction | 19 months
Evaluation of the feasibility of the autologous MSC intracavernous injection protocol by the quality of the bone marrow samples | 19 months
Evaluation of the feasibility of the autologous MSC intracavernous injection protocol by the quality of the cell culture of the marrow of diabetic patients | 19 months
Evaluation of the feasibility of the autologous MSC intracavernous injection protocol by the cell transport delay (between preparation and injection) | 19 months
Evaluation of the feasibility of the autologous MSC intracavernous injection protocol by the patient recruitment rate calculated by the ratio between the number of participants and the number of eligible patients | 19 months
Evaluation of the feasibility of the autologous MSC intracavernous injection protocol by the Injection rate actually achieved | 19 months